CLINICAL TRIAL: NCT03521921
Title: GIse Registry Of Transcatheter Treatment of Mitral Valve regurgitaTiOn (GIOTTO)
Acronym: GIOTTO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Francesco Bedogni, Head of Cardiology, IRCCS Policlinico S. Donato
Other Study IDs: GISE/01/2014/GIOTTO
Record Dates: First submitted 2018-02-05; First posted 2018-05-11 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Mitraclip — Edge-to edge mitral valve repair

SUMMARY:
The current state of the art management of severe mitral regurgitation is surgical mitral valve repair, either with open chest surgery or mini-thoracotomy. However, standard surgical approaches requiring cardiopulmonary bypass are suitable for patients with low or moderate surgical risk, thus many patients are denied surgery because of unfavorable risk-benefit balance. The EuroHeart Surveyconducted by the ESC showed that one half of patients with severe mitral regurgitation were denied surgical treatment because they were felt to be at too high risk for surgery by the referring physician. Such patients are usually elderly and have co-morbidities. Thus, there is a need for novel devices enabling interventional cardiologists and cardiothoracic surgeons to perform mitral repair in a minimally-invasive fashion and possibly without cardiopulmonary bypass. The landmark EVEREST II trial randomized 279 patients with grade 3/4 MR in a 2:1 fashion to MitraClip® or surgical repair/replacement showing a lower major adverse event rate at 30-days in the MitraClip® group (15.0% vs. 48%; superiority p<0.001), mainly driven by the need for blood transfusion with surgery, and the primary efficacy endpoint of freedom from the combined outcome of death, new surgery for mitral valve dysfunction or the occurrence of >2+ MR was achieved in 55% vs. 73% (non-inferiority p=0.007). However, this study has included a highly selected patient cohort in which patients with significant surgical risk have been excluded. More recently, Multinational (ACCESS-EU, EVEREST-High Risk) and national registries (TRAMI, SWISS) have shown safety and efficacy in the real world experience. Patients currently treated are high risk, elderly, with comorbidities and mainly affected by FMR. There is need for an Italian registry, since Italy has produced the second largest volume of transcathetermitral procedures in the world after Germany. The present registry is designed to collect real world clinical data on early and long-term outcomes following percutaneous mitral regurgitation therapy in consecutive patients undergoing transcatheter procedures in Hospitals linked to the GISE database.

DETAILED DESCRIPTION:
The main objective is to achieve demographic and outcome data and identify predictors of clinical success, according to real-world Italian data. In addition the registry is designed to obtain health economic data to support reimbursement strategies in Italy. The study is focusing on MITRACLIP therapy since this is the leading method for treatment currently in Italy.

All consecutive patients undergone/ undergoing a transcatheter mitral valve repair, with Mitraclip device, will be enrolled to reach a number of about 1100 patients in about 22 hospitals. Data analysis will be conducted at the end of follow-up period of the last enrolled patient. . Additional data analysis will be done according to specific topics, approved by the scientific board of GISE and or on Ethic Committees requests. The population of the study is patients undergoing/undergone a transcatheter mitral valve repair procedure in hospitals linked to the GISE network. More specifically Patients from the investigators' general Mitraclip treatment patient population will be eligible to be enrolled in this Registry. Patients should meet all the inclusion criteria and none of the exclusion criteria. Retrospective enrolments are allowed if available data are in line with the Study requirements and the patients can give their consent to be enrolled in the study informed consent process.

Follow-up visit will be performed at 30 days, 1 year and up to 5 years after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are eligible for Mitraclip device according to current national and international guidelines (and their future revisions) and per investigator evaluation;
* Patients who are willing and capable of providing informed consent, participating in all Follow-ups associated with this clinical investigation at an approved clinical investigational center;

More specifically patients inclusion criteria are in line with the indications for use detailed in the IFU in particular, patients have to meet the following inclusions criteria

1. Symptomatic severe (4+) MR, or 3+ MR and NYHA > II.
2. Mitral valve anatomy should be suitable for MitraClip.
3. Signed (by subject or legal representative) and dated approved subject informed consent form prior to any study related data collection.

Exclusion Criteria:

* Valve anatomy is unsuitable for MitraClip therapy as per the indication in the Mitraclip IFU
* Currently participating in the study of an investigational drug or device
* The subject is unable or not willing to complete follow-up visits and examination for the duration of the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any subject who already received or deemed suitable and selected by the site to receive the Mitraclip treatment, in accordance with all applicable device Instructions For Use, should be considered for entry into this study.
  Eligibility will be documented on the inclusion/exclusion criteria sheet. Subjects who meet the eligibility criteria and have signed and dated the Informed Consent Form and actually undergone / undergo a Mitraclip implant procedure are considered enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2016-02-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2025-09-09 (Estimated)

PRIMARY OUTCOMES:
Mortality | From index procedure up to 5 years
  cardiovascular and non-cardiovascular death events with specificed cause.

SECONDARY OUTCOMES:
MACCE | From index procedure up to 5 years
  cardiovascular and cerebrovascular major adverse events.
Reduction of MR | Within 7 days after procedure and 1 year and up to 5 years.
  Reduction of MR evaluated with a scale 1 to 4

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Bedogni, Dr., Principal Investigator — IRCCS Policlinico S. Donato
Locations (20):
- Italy (20):
  - IRCCS Policlinico San Donato, San Donato Milanese, Milan
  - ASST Papa Giovanni XXIII, Bergamo
  - Fondazione Poliambulanza, Brescia
  - Spedali Civili, Brescia
  - Pineta Grande, Castel Volturno
  - Ospedale Ferrarotto, Catania
  - Cardiologia Università Magna Graecia, Catanzaro
  - Maria Cecilia Hospital, Cotignola
  - Ospdale dell'Angelo ULSS12 Veneziana, Mestre
  - Centro Cardiologico Monzino, Milan
  - Ospedale San Raffaele - Cardiochirurgia, Milan
  - Ospedale San Raffaele - Emodinamica, Milan
  - AORN Dei Colli "V. Monaldi - Cardiologia Interventistica, Napoli
  - AORN dei Colli "V. Monaldi" - Emodinamica, Napoli
  - UOC cardiologia Università di Padova, Padua
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - IRCCS Humanitas, Rozzano
  - AOU San Giovanni di Dio e Ruggi D'Aragona, Salerno

IPD SHARING:
Plan to Share IPD: No
The data will be reviewed by a Data Safety and Monitoring Board.
  The Data Safety and Monitoring Board will be also responsible for:
  * Determining whether information collected are sufficient to address the objectives
  * Recommending modifications to the statistical analysis plan to address additional research questions based on review of the data